CLINICAL TRIAL: NCT03723109
Title: Airway Management and Safety Aspects During Target Controlled Infusion (TCI) Compared to Rapid Sequence Induction (RSI) of Anesthesia in Non-cardiac Surgery
Brief Title: Airway Management During TCI vs RSI Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Myrberg, Senior lecturer, MD PhD, Umeå University
Other Study IDs: 2016/361-31 IV
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Adverse Effect; Anesthesia; Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Induction of anesthesia — Standardized TCI and RSI anesthesia induction
  Other Names: Anesthesia induction

SUMMARY:
The aims of this observational study is to evaluate and compare feasibility of airway management during standardized TCI and RSI anesthesia induction.

DETAILED DESCRIPTION:
The aims of this study are to evaluate and compare feasibility of airway management and risk for desaturation during standardized target controlled infusion (TCI) and rapid sequence induction (RSI) of anesthesia. A conventional way to induce anesthesia, i.e. manual injection of anesthetics, may be more accurate and predictable compared to dosing regimes based on complex mathematical algorithms used in TCI-systems. In addition, today many different models are presented and there is no consensus which kind of TCI-algorithm should be used universally. Moreover, dosing algorithms are most complex and challenging in underweight and morbid obesity. There are many publications on this field, but no data of feasibility of airway management can be found. Indeed, RSI induction is traditionally blamed to be risky and not recommended as a first choice.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* BMI < 35 kg/m2
* preoperative assessment accepted by consultant anesthesiologist
* scheduled for breast cancer surgery, endocrinological surgery (thyroid, parathyroid) or minor general abdominal surgery.

Exclusion Criteria:

* not signed consent
* instable angina pectoris
* severe bronchial asthma
* severe chronic obstructive pulmonary disease
* dementia
* severe heart valve disease
* severe renal failure
* body mass index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cohort, electively scheduled for breast cancer surgery, endocrinological surgery (thyroid, parathyroid) and minor general abdominal surgery.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Safety time for apnea | 10min
  measurement of length of period for apnea during TCI and RSI induction by a timer

SECONDARY OUTCOMES:
Duration of spontaneous breathing | 10min
  measurement of duration of spontaneous breathing during TCI and RSI induction by a timer

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Myrberg, MD PhD, Principal Investigator — Umea University, senior lecturer
Locations (1):
- Sunderby teaching hospital, Luleå, Sweden

IPD SHARING:
Plan to Share IPD: No